CLINICAL TRIAL: NCT02532452
Title: Third Party Viral Specific T-cells (VSTs) for Treatment of Viral Infections in Immunocompromised Patients
Brief Title: Third Party Viral Specific T-cells (VSTs)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-4184
Record Dates: First submitted 2015-08-21; First posted 2015-08-25 (Estimated); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Viral Infection; Viral Reactivation; Infection in an Immunocompromised Host
Keywords: Epstein-Barr Virus (EBV); Adenovirus (ADV); Cytomegalovirus (CMV); T-Cells; Donor; BK virus (BKV)
MeSH Terms: conditions — Virus Diseases; Epstein-Barr Virus Infections; Adenoviridae Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Viral Specific VST Infusion (Experimental): 3rd party VST infusion
  Interventions: Biological: Viral Specific VST Infusion

INTERVENTIONS:
Biological: Viral Specific VST Infusion — VSTs will be infused into immunocompromised patients with evidence of viral infection or reactivation defined as any of the following:
  * Blood adenovirus PCR ≥ 1,000
  * Blood CMV PCR ≥ 500
  * Blood EBV PCR ≥ 9,000
  * Plasma BKV PCR >1,000
  * Plasma JC Virus PCR > 1,000
  * Evidence of invasive adenovirus infection or disease, defined as the presence of adenoviral positivity by PCR or culture in one or more sites
  * Evidence of invasive CMV infection, eg pneumonitis, retinitis, colitis
  * Evidence of invasive EBV disease/infection, EBV-associated lymphoproliferation (EBV-LPD) defined as proven EBV-LPD by biopsy or probable EBV-LPD defined as an elevated EBV DNA level in the blood associated with clinical symptoms (adenopathy or fever or masses on imaging) but without biopsy confirmation, or EBV-associated malignancies
  * Evidence of symptomatic BK virus infection, which may include symptomatic hemorrhagic cystitis, or BK nephropathy
  * Evidence of PML or other CNS infection due to JC virus

SUMMARY:
The purpose of this study is to demonstrate that viral specific T-cells (a type of white blood cell) can be generated from an unrelated donor and given safely to patients with viral infections.

DETAILED DESCRIPTION:
Viral reactivation and infection is a major cause of morbidity in immunocompromised patients (including HSCT recipients). In this study we will draw blood from unrelated (third party) donors and use the blood to generate viral specific T-cells (VSTs) with specificity for Epstein-Barr virus (EBV), cytomegalovirus (CMV), adenovirus (ADV), BK virus (BKV), and JC Virus. The VSTs will be infused into immunocompromised children with specific viral infections (EBV, CMV, ADV, BKV , or JC virus). Cells will be selected for infusion based on the recipient's HLA type and the viral specificity of the cells.

ELIGIBILITY:
Inclusion Criteria:

* Immunocompromised patient with evidence of viral infection or reactivation
* Age >1 day
* Recipients who have had a stem cell transplant must be at least 21 days after stem cell infusion
* Clinical status must allow tapering of steroids to < 0.5mg/kg prednisone or other steroid equivalent
* Must be able to receive CTL infusion in Cincinnati
* Informed consent obtained by PI or sub-investigator either in person or by phone

Exclusion Criteria:

* Active acute GVHD grades II-IV
* Uncontrolled bacterial or fungal infection
* Uncontrolled relapse of malignancy requiring treatment with chemotherapy
* Infusion of ATG or alemtuzumab within 2 weeks of VST infusion
* Biopsy confirmed acute rejection of solid organ transplant OR empiric treatment of suspected but not confirmed acute rejection of solid organ transplant within the last 30 days

Min Age: 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2015-09-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Successful production of viral specific T-cells | Within 30 days post culture initiation
  Of the patients who had a VST culture initiated, successful production of VST cells is defined as meeting the protocol-defined release criteria.
Percentage of patients who do not have infusional toxicity | Through 30 minutes post infusion
  Patients will be monitored for infusional toxicity
Incidence of GVHD associated with VST infusion | Through 30 days after infusion
  Patients will be monitored for the development of VST associated GVHD

SECONDARY OUTCOMES:
Presence of viral-specific T-cells | At 30 days after infusion
  Presence of viral-specific T-cells in the participant's blood will be assessed by Elispot assay
Viral burden | At 30 days after infusion
  The viral burden will be assessed using the protocol-defined efficacy assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Grimley, MD, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (4):
- United States (4):
  - Akron Children's Hospital, Akron, Ohio
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - The Ohio State University Wexner Medical Center - James Cancer Hospital, Columbus, Ohio

REFERENCES:
- [Derived] Rubinstein JD, Pham G, Sridharan A, Khoury R, Wang YM, Hudda Z, Wilhelm J, Lichtenstein DA, Heyenbruch D, Cancelas JA, Davies SM, Lutzko C, Grimley MS. Outcomes with third-party virus-specific T cells after the use of single-antigen cell lines to predict HLA restriction. Blood Adv. 2025 Dec 23;9(24):6305-6313. doi: 10.1182/bloodadvances.2025017097. PMID 40991376
- [Derived] Galletta TJ, Lane A, Lutzko C, Leemhuis T, Cancelas JA, Khoury R, Wang YM, Hanley PJ, Keller MD, Bollard CM, Davies SM, Grimley MS, Rubinstein JD. Third-Party and Patient-Specific Donor-Derived Virus-Specific T Cells Demonstrate Similar Efficacy and Safety for Management of Viral Infections after Hematopoietic Stem Cell Transplantation in Children and Young Adults. Transplant Cell Ther. 2023 May;29(5):305-310. doi: 10.1016/j.jtct.2023.01.027. Epub 2023 Feb 3. PMID 36736781
- [Derived] Rubinstein JD, Zhu X, Leemhuis T, Pham G, Ray L, Emberesh S, Jodele S, Thomas S, Cancelas JA, Bollard CM, Hanley PJ, Keller MD, Grimley O, Clark D, Clark T, Lindestam Arlehamn CS, Sette A, Davies SM, Nelson AS, Grimley MS, Lutzko C. Virus-specific T cells for adenovirus infection after stem cell transplantation are highly effective and class II HLA restricted. Blood Adv. 2021 Sep 14;5(17):3309-3321. doi: 10.1182/bloodadvances.2021004456. PMID 34473237
- [Derived] Nelson AS, Heyenbruch D, Rubinstein JD, Sabulski A, Jodele S, Thomas S, Lutzko C, Zhu X, Leemhuis T, Cancelas JA, Keller M, Bollard CM, Hanley PJ, Davies SM, Grimley MS. Virus-specific T-cell therapy to treat BK polyomavirus infection in bone marrow and solid organ transplant recipients. Blood Adv. 2020 Nov 24;4(22):5745-5754. doi: 10.1182/bloodadvances.2020003073. PMID 33216887